CLINICAL TRIAL: NCT05966337
Title: Effects of Non-invasive Ventilation With Different Modalities in Patients Undergoing Heart Surgery: a Randomized Controlled Clinical Trial
Brief Title: Effects of Non-invasive Ventilation in Patients Undergoing Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Collaborators: Universidade Estadual da Paraiba (Other)
Responsible Party: Principal Investigator, Patri-cia Angelica de Miranda Silva Nogueira, Head professor of physiotherapy course and pós-graduate course., Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERAECR12023; 65600722.1.0000.5187 (Other: CAAE)
Record Dates: First submitted 2023-06-08; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Cardiac Surgical Procedures; Continuous Positive Airway Pressure; BIPAP Biphasic Intermittent Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Pacients will be divided into 3 groups (CPAP group - CPAP + usual physical therapy care, BiPAP group - BiPAP + usual physical therapy care, and Control group - usual physical therapy care) in a 1:1 allocation ratio. Control group will receive the usual physiotherapy treatment, as kinesiotherapy protocol. Treatment will be administered twice a day, starting in the ICU and progressing to the ward. In the CPAP group, nasal CPAP at 10cmH2O will be administered for 1 hour, twice a day, using an approved device. In BiPAP group, nasal BiPAP with IPAP of 13cmH2O and EPAP of 8cmH2O will be administered for 1 hour, twice a day, using an approved device. The NIV sessions will be conducted during the 5 days of hospitalization, both in the ICU and the ward. After the fifth day, patients in intervention groups will undergo reassessment using the same assessment instruments as before.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a single-center, randomized, controlled, double-blind clinical trial, in which participants and outcome evaluators were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group 1 (usual care) (Active Comparator): Patients undergo physiotherapy treatment twice daily, transitioning from the ICU to the ward. The treatment plan spans several days, starting on the first postoperative day after ICU discharge. In the ICU, Day 1 includes diaphragmatic breathing exercises, coughing stimulus, upper limb exercises (shoulder flexion/extension, abduction), and lower limb exercises (thigh flexion, dorsiflexion/plantarflexion). Day 2 involves diaphragmatic breathing, coughing stimulus, upper limb exercises, lower limb exercises, cycling for 3 minutes, and respiratory device exercises. Upon moving to the ward on Day 3, patients perform diaphragmatic breathing, coughing stimulus, upper limb exercises, lower limb exercises, and a 5-minute walk. Day 4 focuses on diaphragmatic breathing, coughing stimulus, and a 10-minute walk. Finally, on Day 5, patients engage in diaphragmatic breathing, coughing stimulus, and a 15-minute walk.
  Interventions: Procedure: Usual care in phisicaltherapy
- Intervention group 2 (CPAP) (Experimental): They will be submitted to the same care as the control group, adding NIV with nasal CPAP 10cmH2O for 1 hour using device and brand approved by ANVISA, during the 5 days of hospitalization, both in the ICU and in the ward. The frequency of the sessions will be two (2) per day, in the morning and in the afternoon. Flexibility of time for carrying out the procedure is also planned, since in a hospital environment the patient can often undergo exams, other behaviors that may make it difficult to apply the protocol at the initially scheduled time. After the fifth day, the patient will be reassessed with the same instruments reported.
  Interventions: Procedure: CPAP; Procedure: Usual care in phisicaltherapy
- Intervention group 2 (BIPAP): (Experimental): They will undergo the same care as the control group, adding NIV with nasal BIPAP with IPAP of 13cmH2O and EPAP 8 cmH2O for 1 hour, using equipment and brand approved by ANVISA, during the 5 days of hospitalization, both in the ICU and in the ward . The frequency of the sessions will be two (2) per day, in the morning and in the afternoon. Flexibility of time for carrying out the procedure is also planned, since in a hospital environment the patient can often undergo exams, other behaviors that may make it difficult to apply the protocol at the initially scheduled time. After the fifth day, the patient will be reassessed with the same instruments reported.
  Interventions: Procedure: BIPAP; Procedure: Usual care in phisicaltherapy

INTERVENTIONS:
Procedure: CPAP — Use of non-invasive ventilation in patients in group 2 with CPAP.
  Arms: Intervention group 2 (CPAP)
Procedure: BIPAP — Use of non-invasive ventilation in patients in group 3 with BIPAP.
  Arms: Intervention group 2 (BIPAP):
Procedure: Usual care in phisicaltherapy — Patients undergoing usual physiotherapy treatment, consisting of a kinesiotherapy protocol

SUMMARY:
The goal of this randomized controlled clinical trial is to compare effects of non-invasive ventilation with different modalities (notably CPAP and BIPAP) in patients undergoing heart surgery. The main question[s] it aims to answer are:

* Which NIV ventilation mode is most effective in cardiac surgery patients?
* Is there a big difference between conventional physiotherapy treatment and the use of NIV in these patients? Participants will be submited in the intervention will initially take place in the specific ward that receives patients in the postoperative period of cardiac surgery. Participants will be recruited after the patient is hospitalized the day before the surgery, during which time he will undergo a preoperative evaluation based on the study criteria. On that first day, the evaluation will consist of anamnesis and physical examination, focusing on the history of cardiac disorders, followed by measurements inherent to the protocol. Manovacuometry, chest X-ray, quality of life questionnaire, walk test and spirometry. The evaluation can be carried out in two stages, if there are other demands for the patient during his hospitalization.

Researchers will compare three groups: 1 - cpap group - CPAP + usual physical therapy care, 2 - Bipap group - BIPAP + usual physical therapy care and 3 - Control - usual physical therapy care), in the 1:1 allocation ratio and superiority. to see if the effects of non-invasive ventilation with different modalities in patients undergoing cardiac surgery demonstrates some superior way in clinical practice. The observed outcomes will be: evaluation between NIV modalities, spirometry, lung capacity and vital signs. Secondary outcomes included are degree of satisfaction with the global perception of change scale, and MIF - functional independence measure and blood gas parameters.

DETAILED DESCRIPTION:
The study protocol was conducted following the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) checklist. This is a single-center, randomized, controlled, double-blind clinical trial, in which participants and outcome evaluators were blinded. The study will be submitted to the ethics committee of the State University of Paraíba (UEPB) and carried out in accordance with the Declaration of Helsinki. All participants must provide written informed consent prior to participation, and the study will be registered on the CLINICALTRIALS platform. All participants must provide written informed consent prior to participation. Participants will be divided into three groups (cpap group - CPAP + usual physical therapy care, bipap group - BIPAP + usual physical therapy care and control group - usual physical therapy care), in a 1:1 allocation ratio and superiority.

The project will be carried out at Hospital João XXIII in the city of Campina Grande, Paraíba, Brazil. It is a private hospital affiliated with the SUS network, a reference in cardiology and especially in cardiac surgery for a good part of the state and surrounding states. It presents in its weekly program an average of 8 cardiac surgeries. The evaluation and intervention will take place in the ICU and ward.

Post-randomization exclusion criteria: In case of undertaking any treatment in the hospital environment that contraindicates participation in the study (pacemaker implantation, pneumothorax requiring chest drainage, for example), death or other decompensations not related to the research and return to the ICU .

Criteria for non-adherence to the intervention: Patient who does not perform 3 or more sessions in a row, who withdrew from participating in the study and who has some cardiac arrhythmia (atrial fibrillation, bradycardia) for two sessions even after medication used to contain and pause for rest.

Non-retention criteria: Patient who does not perform one of the reassessments. Professional eligibility criteria: Hospital staff physiotherapists and physiotherapy students with previous training in the research protocol.

Procedures for Conducting the Research The purpose of this project is to carry out a randomized clinical trial and verify the effectiveness of NIV compared to conventional physiotherapy in terms of the rate of pulmonary complications in patients undergoing cardiac surgery in a chosen hospital in the city of Campina Grande, Paraíba.

Thus, there will be a partnership with the Núcleo de Tecnologia Estratégicas em Saúde (NUTES) of the State University of Paraíba (UEPB) through the biomedical computing laboratory for the development of research aimed at the remote monitoring of health data through smartwatches and other devices that comply with international standardization norms for interoperability between health technologies. NUTES already collaborates with UFRN in several scientific and technological cooperation researches, so that the co-supervisor of the project, Prof Paulo Eduardo Barbosa made the strategic partnership possible, according to the attached document. NUTES' participation in this project will take place through the feasibility of remote monitoring technology via Smartwatch and the introduction of data collected on a specific platform.

For a better understanding and operationalization of the research, it was divided into 5 phases.

1. st Phase: Documentary Survey and Consent At first, there was initial contact with the aforementioned hospital institution for consent to the research. At the same time, a documentary and systematic study on the subject was instituted, in order to base the research and identify possible indices and/or parameters that would add to the research in order to make it viable and absolutely realistic.
2. nd Phase: Search and profile of NIV and Smartwatch devices Non-invasive ventilation (NIV) will be performed both in the ICU environment and in the ward for the intervention group. A BIPAP will be made available and a CPAP for the respective groups. The interface chosen will be the nasal mask, aiming at greater patient comfort. Thus, we will choose properly calibrated NIV devices on the market that provide better adaptation to patients.

   All the main information about users can be entered into the platform, such as gender, age, other illnesses, use of medication, and some special situations that can be verified in practice, in addition to information that may come from the monitoring carried out by the smartwatch on patients in the moment of data collection during NIV application. Thus, data from the patient's medical record will also be used. A large volume of data can be entered into the platform and used to generate a profile of cardiac patients selected for the survey. The smartwatch used will be from the Garmin brand and available for capturing Sao2 and VO2.

   The main functionalities of the Dashboard comprise the visualization of the data of the surgical patients submitted to NIV in the initial screen in a computer, being able to apply filters according to the interest of the researcher.
3. rd Phase: Technical Study and applied tests

   This project is interested in three major aspects: the use of non-invasive ventilation in heart patients undergoing cardiac surgery; the automation of data collection using the smartwatch, making it practical, simple, accessible technology in order to become a predictor of safe discharge for these patients; finally, a survey of a large volume of data (verified in the analysis profile of the patients) that can generate subsidies for carrying out research and contribute to the increase of studies in the area of cardiopulmonary physiotherapy on technological bases.
4. th Phase: Pilot Study - Practice After that, the surgeries will begin and the collection will consist of 6 patients, thus defining the beginning of the pilot study. Upon being notified of the weekly surgical schedule, the researcher in charge will randomize the patients. This register will contain the complete identification of the patient, type of surgery to which he will be submitted and the pathology.

   Thus, as the patients leave the surgical center and go to the ICU, they will follow the protocol so that the treatment due to the group to which the patient is allocated on the day after the surgery begins.

   It should be noted that the pilot study should only be started after approval by CEP.

   After completion of the pilot study, there will be an evaluation of the entire protocol so that possible flaws can be corrected before definitive collection.
5. th Phase: Data collection It will consist of collecting data from patients in the post-randomization intervention and allocation of patients to a group, following the procedures of the protocol.

ELIGIBILITY:
Inclusion Criteria: Patients undergoing cardiac surgery

* aged over 18 years
* stable from the hemodynamic point of view (controlled blood pressure, normocardic
* conscious and oriented and cooperative4
* without medical restrictions for carrying out the treatment

Exclusion Criteria:

* Presence of uncontrolled cardiac arrhythmias (Examples: total atrioventricular block, type 2 2nd degree atrioventricular block, atrial fibrillation, sustained ventricular tachycardia)
* previous neuromuscular disease
* labyrinthitis and some orthopedic/skeletal muscle restriction.
* Unstable angina, stage 3 SAH (SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg at rest), HR > 120 bpm at rest, systemic arterial hypotension with clinical repercussions (SBP ≤ 90 mmHg and/or DBP ≤ 60 mmHg),(),
* aortic dissection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function | Day 1 and day 5
  All participants will undergo an evaluation by a CONTEC model spirometer (SPB80b, CHINA) to verify lung volumes and capacities. At least three tests will be performed, with a variation of less than 5% and the highest value obtained in one of the tests will be compared with the predicted values of pulmonary function parameters for the Brazilian population. FEV1 and FVC will be assessed. The predicted values will be calculated using the reference values (PEREIRA et al., 2007).
Length of hospital stay | The length of hospital stay will be assessed and reported as the number of days from admission to discharge, measured up to 2 weeks after the date of randomization.
  Absolute number of days of hospitalization up to 2 weeks after the date of randomization.
Presence of lung complications | From the date of randomization to the date of the first documented progression or the date of death from any cause, whichever occurs first, measured up to 2 weeks after the date of hospital discharge.
  assessment of the occurrence or absence of any complications related to the lungs during the hospitalization period.cause, whichever occurs first, measured up to 2 weeks

SECONDARY OUTCOMES:
Score of the Minnesota Living with Heart Failure Questionnaire (MLHFQ) in Portuguese version | Day 1 and Day 5
  The Portuguese version of the MLHFQ will be used to assess the patient's quality of life. The questionnaire provides a final score as a metric, and the change in score over the treatment period will be evaluated. The MLHFQ score is a measure of health-related quality of life in patients with heart failure. The higher the score, the greater the negative impact of heart failure on the patient's quality of life. A score of 0 indicates that the patient has no limitations or problems related to heart failure, while a score of 105 indicates a maximum limitation or problem in all areas assessed by the questionnaire.
Funcional capacity | Day 1 and Day 5
  The TUG test will be performed to assess functional capacity. The patient will start from a sitting position, walk quickly for 3 meters, turn 180 degrees, and return to the chair. The time taken, measured from standing up to completely leaning the trunk against the chair, will be recorded. Time values below 10 seconds indicate maximum functionality, 10 to 19 seconds indicate functional independence, 20 seconds and above indicate some functional limitation, and 30 seconds and above indicate significant functional limitation.
The global perception of change scale | Day 1 and Day 5
  The GPCS is a self-report tool that assesses an individual's perception of change in a specific domain. It uses Likert-scale items ranging from "a very great deal worse/less" to "a very great deal better/more" to capture subjective information about perceived change.
The functional independence measure (MIF) | Day 1 and Day 5
  The MIF questionnaire will be administered preoperatively and on the sixth day to assess functional independence.
pO2 (partial pressure of oxygen) | Days 1 and 2.
  Partial pressure of oxygen (PO2) is a key physiological parameter that measures the pressure exerted solely by oxygen molecules in a mixture of gases, such as air or blood. It is an important indicator of the oxygen-carrying capacity and oxygen exchange efficiency in the respiratory system (ROCA et al. 2020). PO2 will be measured in millimeters of mercury (mmHg) (BAI, et al. 2020)
pCO2 (partial pressure of carbon dioxide) | Days 1 and 2.
  Partial pressure of carbon dioxide (pCO2) is a fundamental physiological parameter that measures the pressure exerted solely by carbon dioxide molecules in a mixture of gases, such as air or blood. It plays a crucial role in the regulation of acid-base balance and respiratory function.
  The unit of measurement for pCO2 will be expressed in millimeters of mercury (mmHg).(RODRIGUEZ, 2006)
HCO3 (bicarbonate) | Days 1 and 2.
  Bicarbonate (HCO3) is an important physiological parameter that measures the concentration of bicarbonate ions in the blood. It is a vital component of the body's acid-base balance and plays a crucial role in maintaining the pH of the blood within a normal range.
  The unit of measurement for bicarbonate will be expressed in milliequivalents per liter (mEq/L) (CHUA, 2011).
Arterial Oxygen Saturation (SaO2) | Days 1 and 2.
  Arterial Oxygen Saturation (SaO2) is a critical physiological parameter that measures the percentage of hemoglobin in arterial blood that is bound with oxygen. It reflects the efficiency of oxygen transport from the lungs to the body's tissues.
  The unit of measurement for SaO2 is typically expressed as a percentage (%). (CASTRO, et al, 2022)
Base Excess (BE) | Days 1 and 2.
  Base Excess (BE) is a significant physiological parameter that measures the amount of excess or deficit of base (bicarbonate) in the blood, indicating the body's acid-base balance. It quantifies the deviation of the blood's buffering capacity from the normal range, which helps in assessing the metabolic component of acid-base disturbances.
  The unit of measurement for Base Excess will be expressed in milliequivalents per liter (mEq/L) (CASTRO, et al, 2022)

OTHER OUTCOMES:
Duration of Cardiopulmonary Bypass | Day 1
  The duration of cardiopulmonary bypass during the cardiac surgery. • Unit of Measure: minutes
Type of Surgery | Day 1
  The specific type of cardiac surgery performed. • Unit of Measure: N/A (Categorical Variable)
Personal History | Day 1
  Relevant information about the patient's personal medical history. • Unit of Measure: N/A (Categorical Variable)
Preoperative Ejection Fraction | Day 1
  The percentage of preoperative cardiac ejection fraction.• Unit of Measure: percentage (%)
Previous Respiratory Complications | Day 1
  Indication of the presence or absence of previous respiratory complications. • Unit of Measure: N/A (Categorical Variable)
Body Mass Index (BMI) | Day 1
  The patient's body mass index, calculated as weight (in kg) divided by the square of height (in meters). Unit of Measure: N/A (Calculated from weight and height)
Gender | Day 1
  The patient's gender (male or female). Unit of Measure: N/A (Categorical Variable)
Age | Day 1
  The patient's age in years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital João XXIII, Campina Grande, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hossen A, Jaju D, Al-Abri M, Al-Sabti H, Mukaddirov M, Hassan M, Al-Hashmi K. Investigation of heart rate variability of patients undergoing coronary artery bypass grafting (CABG). Technol Health Care. 2017;25(2):197-210. doi: 10.3233/THC-161260. PMID 28387685
- [Background] Du H, Newton PJ, Salamonson Y, Carrieri-Kohlman VL, Davidson PM. A review of the six-minute walk test: its implication as a self-administered assessment tool. Eur J Cardiovasc Nurs. 2009 Mar;8(1):2-8. doi: 10.1016/j.ejcnurse.2008.07.001. Epub 2008 Aug 9. PMID 18694656
- [Background] Shakouri SK, Salekzamani Y, Taghizadieh A, Sabbagh-Jadid H, Soleymani J, Sahebi L, Sahebi R. Effect of respiratory rehabilitation before open cardiac surgery on respiratory function: a randomized clinical trial. J Cardiovasc Thorac Res. 2015;7(1):13-7. doi: 10.15171/jcvtr.2015.03. Epub 2015 Mar 29. PMID 25859310
- [Background] Valkenet K, de Heer F, Backx FJ, Trappenburg JC, Hulzebos EH, Kwant S, van Herwerden LA, van de Port IG. Effect of inspiratory muscle training before cardiac surgery in routine care. Phys Ther. 2013 May;93(5):611-9. doi: 10.2522/ptj.20110475. Epub 2013 Jan 3. PMID 23288909
- [Background] Dos Santos TD, Pereira SN, Portela LOC, Cardoso DM, Lago PD, Dos Santos Guarda N, Moresco RN, Pereira MB, de Albuquerque IM. Moderate-to-high intensity inspiratory muscle training improves the effects of combined training on exercise capacity in patients after coronary artery bypass graft surgery: A randomized clinical trial. Int J Cardiol. 2019 Mar 15;279:40-46. doi: 10.1016/j.ijcard.2018.12.013. Epub 2018 Dec 10. PMID 30581100
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Carvalho VO, Guimaraes GV, Carrara D, Bacal F, Bocchi EA. Validation of the Portuguese version of the Minnesota Living with Heart Failure Questionnaire. Arq Bras Cardiol. 2009 Jul;93(1):39-44. doi: 10.1590/s0066-782x2009000700008. English, Portuguese, Spanish. PMID 19838469
- [Background] 8. Vieira WO, Barbosa LK, Bezerra AS, et al. Test timed up and go and its correlation with age and functional exercise capacity in asymptomatic women. Fisioterapia em Movimento. 2017;30(3):463-471. doi:10.1590/1980-5918.030.003.AO04.
- [Background] Bretan O, Silva Junior JE, Ribeiro OR, Corrente JE. Risk of falling among elderly persons living in the community: assessment by the Timed up and go test. Braz J Otorhinolaryngol. 2013 Jan-Feb;79(1):18-21. doi: 10.5935/1808-8694.20130004. PMID 23503902
- [Background] Behlouli H, Feldman DE, Ducharme A, Frenette M, Giannetti N, Grondin F, Michel C, Sheppard R, Pilote L. Identifying relative cut-off scores with neural networks for interpretation of the Minnesota Living with Heart Failure questionnaire. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:6242-6. doi: 10.1109/IEMBS.2009.5334659. PMID 19965089
- [Background] Bai C, Chotirmall SH, Rello J, Alba GA, Ginns LC, Krishnan JA, Rogers R, Bendstrup E, Burgel PR, Chalmers JD, Chua A, Crothers KA, Duggal A, Kim YW, Laffey JG, Luna CM, Niederman MS, Raghu G, Ramirez JA, Riera J, Roca O, Tamae-Kakazu M, Torres A, Watkins RR, Barrecheguren M, Belliato M, Chami HA, Chen R, Cortes-Puentes GA, Delacruz C, Hayes MM, Heunks LMA, Holets SR, Hough CL, Jagpal S, Jeon K, Johkoh T, Lee MM, Liebler J, McElvaney GN, Moskowitz A, Oeckler RA, Ojanguren I, O'Regan A, Pletz MW, Rhee CK, Schultz MJ, Storti E, Strange C, Thomson CC, Torriani FJ, Wang X, Wuyts W, Xu T, Yang D, Zhang Z, Wilson KC. Updated guidance on the management of COVID-19: from an American Thoracic Society/European Respiratory Society coordinated International Task Force (29 July 2020). Eur Respir Rev. 2020 Oct 5;29(157):200287. doi: 10.1183/16000617.0287-2020. Print 2020 Sep 30. PMID 33020069
- [Background] Rodriguez P, Lellouche F, Aboab J, Buisson CB, Brochard L. Transcutaneous arterial carbon dioxide pressure monitoring in critically ill adult patients. Intensive Care Med. 2006 Feb;32(2):309-312. doi: 10.1007/s00134-005-0006-4. Epub 2006 Jan 31. PMID 16450093
- [Background] Chua HR, Schneider A, Bellomo R. Bicarbonate in diabetic ketoacidosis - a systematic review. Ann Intensive Care. 2011 Jul 6;1(1):23. doi: 10.1186/2110-5820-1-23. PMID 21906367
- [Background] Castro D, Patil SM, Zubair M, Keenaghan M. Arterial Blood Gas. 2024 Jan 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK536919/ PMID 30725604
- [Derived] Araujo ER, Bezerra Nogueira ID, E Silva Barbosa PE, Silva Nogueira PAM. Effects of Non-Invasive Ventilation with different modalities in patients undergoing heart surgery: Protocol for a randomized controlled clinical trial. PLoS One. 2024 Jun 18;19(6):e0304569. doi: 10.1371/journal.pone.0304569. eCollection 2024. PMID 38889140